CLINICAL TRIAL: NCT05100953
Title: Application of Physical Activity Counseling Program in Healthy Adult Individuals
Brief Title: Application of Physical Activity Counseling Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Nisa Nur KÖSE, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NKOSE
Record Dates: First submitted 2021-10-05; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Healthy Lifestyle
Keywords: Physical Activity; Quality of Life; Sleep Habits; Depression; Videoconferencing; Telehealth
MeSH Terms: conditions — Motor Activity; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): After informing about the benefits of physical activity at the beginning of the study, physical activity counseling will be applied once a week for two months via videoconference.
  Interventions: Behavioral: Physical Activity Counseling
- Control Group (No Intervention): At the beginning of the study, a one-session briefing will be given on the benefits of physical activity.

INTERVENTIONS:
Behavioral: Physical Activity Counseling — Physical activity counseling will be provided under supervision by the researcher physiotherapist via video conference and an individual physical activity program will be organized weekly for two months.
  Arms: Experimental Group

SUMMARY:
Abstract Implementation of Physical Activity Counseling Program in Healthy Adult Individuals It was planned to investigate the effects of physical activity counseling on physical fitness level, physical activity level, depression level, sleep quality, quality of life and the change in the number of daily steps. 48 healthy adults aged 18-65 years will be included in the study. Participants will be randomized to the experimental group receiving videoconferencing counseling for eight weeks and the control group receiving single-session informational counseling. Participants will be evaluated with online questionnaires and physical fitness tests during the video conference before the study begins, at the end of the first month and at the end of the second month. Online surveys to be applied; PACE Score, Physical Activity Readiness Questionnaire (PAR-Q), Short Form International Physical Activity Questionnaire (IPAQ-SF), Pittsburgh Sleep Quality Index (PUKI), Beck Depression Inventory (BDI), World Health Organization Quality of Life Scale-Short Form ( WHOQOL-BREF) and physical fitness tests; Plank Test, Curl Up Test, Modified Push Up Test and Squat Test. Demographic information of the participants such as age, weight, height will be recorded. In addition, all participants will record their step counts with the pedometer application they download to their phones one week before the study starts and for one week after the study ends.

ELIGIBILITY:
Inclusion Criteria:

* Not having a co-morbid disease that would prevent physical activity
* Having internet access and equipment to make video calls
* Working remotely

Exclusion Criteria:

* Having a diagnosis of any neurodegenerative or chronic disease
* Having significant cardiovascular, neuromuscular or endocrine disorders that limit regular physical activity
* Recent myocardial infarction or other acute cardiac event, unstable angina, uncontrolled cardiac arrhythmias
* In the past 2 months having had Covid 19

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2021-12-20 (Estimated); Study Completion 2022-01-10 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Level | first measurement at the beginning of the study,change at first month, change at second month
  International Physical Activity Questionnaire of Short Form:IPAQ-SF records the last 7 day recall for four intensity levels of physical activity which is vigorous-intensity activity, moderate-intensity activity, walking, and sitting. From IPAQ-SF, data were converted to Metabolic Equivalent minutes per week (MET-min/week) using. Compendium average MET score (Walking = 3.3 METs, Moderate Physical Activity = 4.0 METs and Vigorous Physical Activity = 8.0 METs).
Depression Level | first measurement at the beginning of the study,change at first month, change at second month
  Beck Depression Scale: BDI scores of 0-13 indicate minimal depression, 14-19 (mild depression), 20-28 (moderate depression) and 29-63 (severe depression).
Sleep Quality | first measurement at the beginning of the study,change at first month, change at second month
  Pittsburgh Sleep Quality Index: In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Life Quality | first measurement at the beginning of the study,change at first month, change at second month
  World Health Organization Quality of Life Scale-Short Form: WHOQOL-BREF is a scale for the quality of life assessment developed by the World Health Organization. It is composed by 26 questions graded from 1 to 5.
  Scoring:
  1 to 2.9 - needs improvement 3 to 3.9 - regular 4 to 4.9 - good 5 - very good
  Question 1 asks about the individual's overall perception of quality of life. Results refer to question 1.
Plank Test | first measurement at the beginning of the study,change at first month, change at second month
  The physical fitness of the participants was evaluated with the Plank Test. The plank test is used to measure the strength and endurance of the core area. The duration of stay in the plank position is recorded by the researcher.
Curl Up Test | first measurement at the beginning of the study,change at first month, change at second month
  The physical fitness of the participants was evaluated with the Curl Up Test. The Curl-Up test is used to evaluate the strength and endurance of the abdominal muscles.The number of repetitions made in one minute is recorded.
Modified Push Up Test | first measurement at the beginning of the study,change at first month, change at second month
  The physical fitness of the participants was evaluated with the Modified Push Up Test. The modified Push Up test evaluates chest muscles and upper extremity endurance.The number of modified push-ups performed correctly in succession without rest in 40 seconds is recorded.
Squat Test | first measurement at the beginning of the study,change at first month, change at second month
  The physical fitness of the participants was evaluated with the Squat Test. The squat test evaluates lower extremity muscle endurance.The number of repetitions that the participant can do in one minute is recorded.
Step Counts | first measurement at the beginning of the study, change at second month
  Participants recorded their step counts with a pedometer app they downloaded to their phones.
Body Mass Index | first measurement at the beginning of the study, change at second month
  BMI is calculated by dividing body weight (kg) by the square of the height in meters.

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes